CLINICAL TRIAL: NCT02777619
Title: Pharmacodynamic Interactions of Propofol and Dexmedetomidine on Target-controlled Infusion Intravenous Anesthesia During the Induction
Brief Title: Pharmacodynamic Interactions of Propofol and Dexmedetomidine on Intravenous Anesthesia
Acronym: PIPDIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, Associate Professor, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pharmacodynamic Interactions
Record Dates: First submitted 2016-05-11; First posted 2016-05-19 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-05

CONDITIONS: Pharmacodynamic Interaction
Keywords: Pharmacodynamic; Dexmedetomidine; Propofol; Target-controlled Infusion Intravenous Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Propofol and 0.0ng/ml Dexmedetomidine (Placebo Comparator): Propofol infusion was started to provide an effect-site concentration of 1.0ug/ml after Dexmedetomidine which target plasma concentration is 0.0ng/ml administered for 15min, and increased by 0.2ug/ml until the patient's consciousness disappears.
  Interventions: Drug: 0.0ng/ml Dexmedetomidine; Drug: Propofol
- Propofol and 0.4ng/ml Dexmedetomidine (Experimental): Propofol infusion was started to provide an effect-site concentration of 1.0ug/ml after Dexmedetomidine which target plasma concentration is 0.4ng/ml administered for 15min, and increased by 0.2ug/ml until the patient's consciousness disappears.
  Interventions: Drug: 0.4ng/ml Dexmedetomidine; Drug: Propofol
- Propofol and 0.6ng/ml Dexmedetomidine (Experimental): Propofol infusion was started to provide an effect-site concentration of 1.0ug/ml after Dexmedetomidine which target plasma concentration is 0.6ng/ml administered for 15min, and increased by 0.2ug/ml until the patient's consciousness disappears.
  Interventions: Drug: 0.6ng/ml Dexmedetomidine; Drug: Propofol
- Propofol and 0.8ng/ml Dexmedetomidine (Experimental): Propofol infusion was started to provide an effect-site concentration of 1.0ug/ml after Dexmedetomidine which target plasma concentration is 0.8ng/ml administered for 15min, and increased by 0.2ug/ml until the patient's consciousness disappears.
  Interventions: Drug: 0.8ng/ml Dexmedetomidine; Drug: Propofol

INTERVENTIONS:
Drug: 0.0ng/ml Dexmedetomidine — Dexmedetomidine target plasma concentration is 0.0ng/ml
  Arms: Propofol and 0.0ng/ml Dexmedetomidine
Drug: 0.4ng/ml Dexmedetomidine — Dexmedetomidine target plasma concentration is 0.4ng/ml
  Arms: Propofol and 0.4ng/ml Dexmedetomidine
Drug: 0.6ng/ml Dexmedetomidine — Dexmedetomidine target plasma concentration is 0.6ng/ml
  Arms: Propofol and 0.6ng/ml Dexmedetomidine
Drug: 0.8ng/ml Dexmedetomidine — Dexmedetomidine target plasma concentration is 0.8ng/ml
  Arms: Propofol and 0.8ng/ml Dexmedetomidine
Drug: Propofol

SUMMARY:
The purpose of this study is to determine pharmacodynamic interactions of propofol and dexmedetomidine,exploring the effect of dexmedetomidine on propofol unconsciousness median effective concentration (EC50).

DETAILED DESCRIPTION:
64 cases were randomly divided into four groups, In each group, dexmedetomidine target plasma concentration are 0, 0.4, 0.6, 0.8 ng/ml. Dexmedetomidine administered 15 min before target controlled infusion of propofol. The propofol infusion was started to provide a target effect-site concentration of 1.0ug/ml, and increased by 0.2ug/ml until loss of consciousness when the effect-site concentration and target concentration equilibrium.

ELIGIBILITY:
Inclusion Criteria:

1. Weight:18≦ BMI≦25
2. Written informed consent from the patient or the relatives of the participating patient.

Exclusion Criteria:

1. A previous history of intolerance to the study drug or related compounds and additives.
2. Existing significant haematological, endocrine, metabolic or gastrointestinal disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The EC50 of propofol for loss of consciousness | within 30 min during the induction of anesthesia
  The aim of the investigators study is to define the optimum target concentration (EC50) of propofol for loss of consciousness with different dexmedetomidine target plasm concentration.

SECONDARY OUTCOMES:
The EC95 of propofol for loss of consciousness | within 30 min during the induction of anesthesia
  The aim of the investigators study is to define the optimum target concentration (EC95) of propofol for loss of consciousness with different dexmedetomidine target plasm concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen Z, Shao DH, Hang LH. Effects of dexmedetomidine on performance of bispectral index as an indicator of loss of consciousness during propofol administration. Swiss Med Wkly. 2013 Mar 14;143:w13762. doi: 10.4414/smw.2013.13762. eCollection 2013. PMID 23519436
- [Background] Hannivoort LN, Eleveld DJ, Proost JH, Reyntjens KM, Absalom AR, Vereecke HE, Struys MM. Development of an Optimized Pharmacokinetic Model of Dexmedetomidine Using Target-controlled Infusion in Healthy Volunteers. Anesthesiology. 2015 Aug;123(2):357-67. doi: 10.1097/ALN.0000000000000740. PMID 26068206